CLINICAL TRIAL: NCT04905498
Title: Developmental Decision Making Study
Brief Title: Promoting Resilience to Food Commercials Decreases Susceptibility to Unhealthy Food Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00003631; 8UG1OD024943-02 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Children were exposed to food commercials without narratives.
  Interventions: Behavioral: Control
- Intervention (Experimental): Children were exposed to narrative statements that were shown and read aloud in between commercials played.
  Interventions: Behavioral: Commercial Advertising Literacy Training

INTERVENTIONS:
Behavioral: Commercial Advertising Literacy Training — Children were shown food commercials and in between those commercials they saw and heard statements such as "These foods won't make you happy" and "Those foods are so unhealthy."
  Arms: Intervention
Behavioral: Control — Children were shown food commercials that were the same length as the other group but did not receive any information about whether the content was truthful.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate how food commercials influence food choices in children and their parents.

DETAILED DESCRIPTION:
The proposed research will investigate food decision-making in youth. Childhood obesity is a risk factor for health issues, thus preventing adverse effects of childhood obesity by promoting healthy eating habits and providing effective interventions are important. Television food commercials advertising calorie-dense and high in salt and sugar foods are known to contribute unhealthy food choices and obesity. Thus the proposed study will examine how the advertising intervention focusing on increasing advertising knowledge and changing affective attitudes toward commercials impacts susceptability to commercials and food decisions in youth.

ELIGIBILITY:
Inclusion Criteria:

* Children had to be between 8-12.9 years old (including 8 year olds, NOT including 13 year olds.
* Had to be able to speak English as their primary language.
* Self-reported normal hearing and vision.

Exclusion Criteria:

* Did not speak English
* Data from children with history of neurological conditions, clinically significant psychopathology, or learning disabilities reported by parents (e.g., Attention Deficit Hyperactivity Disorder, depression) will be excluded.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Bruce, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ha OR, Killian HJ, Davis AM, Lim SL, Bruce JM, Sotos JJ, Nelson SC, Bruce AS. Promoting Resilience to Food Commercials Decreases Susceptibility to Unhealthy Food Decision-Making. Front Psychol. 2020 Dec 2;11:599663. doi: 10.3389/fpsyg.2020.599663. eCollection 2020. PMID 33343472
- See also: Frontiers — http://www.frontiersin.org/articles/10.3389/fpsyg.2020.599663/full
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov/33343472/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 19 | 30
Completed | 18 | 28
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — COVID lockdown | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 19 | 30 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 30 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (1.43) | 10.06 (1.37) | 10.51 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 8 | 13 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 18 | 28
  More than one race | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 30 | 49

OUTCOME MEASURES:

1. Primary Outcome: Food Choice Change
Description: Children rated on a 4-point Likert scale (1-Strong No, 2-No, 3-Yes, 4-Strong Yes) about whether they would choose to eat 60 different foods (30 unhealthy, 30 healthy) on a computer program. Higher values for unhealthy foods represented unhealthier food choices and higher values for healthy foods represented healthier food choices. The mean scores for unhealthy food choices were compared between pre- and post-intervention, and the mean scores for healthy food choices were compared between pre- and post-intervention.
Time Frame: Pre (day 0) and post intervention (day 7-10).
Population: The experimenter assigned children to one of two groups using a random assignment of drawing cell numbers pre-assigned for each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Children were exposed to food commercials without narratives.
  Control: Children were shown food commercials that were the same length as the other group but did not receive any information about whether the content was truthful.
  Taste attributes significantly predicted food decisions for both groups.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 30
score on a scale
  Pre Intervention Unhealthy foods | 3.09 (0.29) | 3.19 (0.37)
  Post Intervention Unhealthy foods | 3.09 (0.37) | 3.07 (0.48)
  Pre Intervention Healthy foods | 2.66 (0.37) | 2.83 (0.39)
  Post Intervention Healthy foods | 2.76 (0.44) | 2.86 (0.36)

2. Primary Outcome: Food Tastiness Change
Description: Children rated on a 4 point Likert scale (1-Very Bad, 2-Bad, 3-Good, 4-Very Good) about how tasty 60 different foods (30 unhealthy, 30 healthy) were on a computer program. A regression coefficient (beta) of food taste was estimated at an individual level by fitting a linear regression model where taste and health ratings predicted food choices for each child. Higher estimated regression coefficients represented higher decision weights of food taste attributes in food choices. The mean estimated regression coefficients were compared between pre- and post-intervention.
Time Frame: Pre (day 0) and post intervention (day 7-10).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 30
beta coefficient
  Pre Intervention | 0.68 (0.22) | 0.75 (0.34)
  Post Intervention | 0.57 (0.28) | 0.59 (0.27)

3. Primary Outcome: Food Health Change
Description: Children rated on a 4 point Likert scale (1-Very Unhealthy, 2-Unhealthy, 3-Healthy, 4-Very Healthy) about how healthy 60 different foods (30 unhealthy, 30 healthy) were on a computer program. A regression coefficient (beta) of food healthiness was estimated at an individual level by fitting a linear regression model where taste and health ratings predicted food choices for each child. Higher estimated regression coefficients represented higher decision weights of food healthiness attributes in food choices. The mean estimated regression coefficients were compared between pre- and post-intervention.
Time Frame: Pre (day 0) and post intervention (day 7-10).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 30
beta coefficient
  Pre Intervention | 0.003 (0.19) | 0.02 (0.24)
  Post Intervention | -0.01 (0.17) | 0.01 (0.16)

4. Secondary Outcome: Level of Self-Control, as Measured by the Self-Control Scale
Description: Children completed the 36-item self-control scale. Each item is rated on a 5-point Likert scale from 1 (not at all like me) to 5 (very much like me). A total score (i.e., 36 response scores were summed) was computed for each child. The total score ranged between 36 (minimum) and 180 (maximum). The higher total score represented higher (better) perceived self-control. No subscales were used.
Time Frame: Children completed this item at the baseline visit (pre intervention).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 19 | 30
scores on a scale | 125.89 (17.01) | 125.00 (14.75)

ADVERSE EVENTS:
Time Frame: 7 to 10 days (between pre and post-intervention)
Groups:
- Control: Children were exposed to food commercials without narratives.
  Control: Children were shown food commercials that were the same length as the other group but did not receive any information about whether the content was truthful.
  No adverse events.
- Intervention: Children were exposed to narrative statements that were shown and read aloud in between commercials played.
  Commercial Advertising Literacy Training: Children were shown food commercials and in between those commercials they saw and heard statements such as "These foods won't make you happy" and "Those foods are so unhealthy."
  No Adverse events.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/30
Other Adverse Events (participants affected / at risk) | 0/19 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT04905498/Prot_SAP_000.pdf